CLINICAL TRIAL: NCT04296669
Title: Stand Out in Class: Reducing Sitting Time in the Classroom Environment
Acronym: SOIC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: Bradford Teaching Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Stacy Clemes, Principle Investigator, Loughborough University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R15-P086
Record Dates: First submitted 2020-02-24; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Sedentary Behavior; Child Behavior; Physical Activity; Obesity; Health Behavior
MeSH Terms: conditions — Sedentary Behavior; Child Behavior; Motor Activity; Obesity; Health Behavior

STUDY DESIGN:
Intervention Model Description: Controlled trial (2 intervention groups)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Full desk allocation (Experimental): All children within this classroom received a sit-stand stand
  Interventions: Device: Ergotron LearnFit Sit-Stand desk
- Partial desk allocation (Experimental): six sit-stand desks were provided in this classroom. Children were rotated between these desks and traditional desks
  Interventions: Device: Ergotron LearnFit Sit-Stand desk
- Control (No Intervention): Traditional classroom furniture was used

INTERVENTIONS:
Device: Ergotron LearnFit Sit-Stand desk — An adjustable sit-stand desk design for children
  Arms: Full desk allocation; Partial desk allocation

SUMMARY:
The primary aim of this study is to examine the effectiveness of incorporating manually adjustable sit-stand desks in the classroom environment of 9-10 year olds in reducing sedentary behaviour at school during a full school year. Secondary aims include evaluating the effects of the intervention on health and learning outcomes as well as comparing the impact of full classroom allocation of sit-stand desks to a classroom of partial sit-stand desk allocation.

DETAILED DESCRIPTION:
Rates of overweight and obesity and related chronic disease risk factors in children have increased worldwide over the past decades. Whilst it is widely acknowledged that regular physical activity provides health benefits, prolonged sedentary behaviour (sitting or reclining) has been shown to adversely affect children's health, independent of the child's physical activity levels. Adverse associations between sedentary behaviour and risk factors for disease, such as obesity, blood pressure, and high levels of cholesterol have been observed in children. In addition, prolonged sedentary behaviour has been linked to reduced cognitive development and academic achievement in children.

Changes in our environment and lifestyle have resulted in children not only becoming less physically active, but also spending unnecessarily long periods of time sitting, particularly in the classroom. Sedentary behaviour is the most prevalent behaviour exhibited by children in developed countries, comprising >65% of waking hours. The impact of unhealthy lifestyle behaviours, such as prolonged sitting, on children's health and development is concerning given the importance of childhood for the establishment of lifestyle behaviours that can track into adulthood.

The long term vision of our research is to re-address the balance between sedentary and non-sedentary (i.e. standing and all forms of physical activity) behaviours by changing environments which are traditionally associated with prolonged periods of sedentary behaviour, such as the school classroom. This study will make environmental changes to the classrooms of Year 5 students (aged 9-10 years) from one school in Bradford, in the UK, through the provision of manually adjustable sit-stand workstations. The primary aim is to compare the effects of this novel strategy using both full desk allocation (one per child) in one classroom and partial desk allocation (six standing desks in a class along with standard desks) in a second classroom on children's classroom sitting and standing time. Comparisons will also be made between the two intervention classrooms in the one school to children's sitting and standing behaviour measured in a control school (following usual practice). Secondary aims include evaluating the effects of the two interventions on time spent in different intensities of physical activity, health, learning and cognitive function outcomes.

This study expands on the success of the nine week pilot study, conducted in 2014, by implementing the intervention over a full academic year, having an additional intervention group, including an extra school for a control group, and including more key outcome measures (blood glucose, self-reported comfort) to better understand the impact of sit-stand desks. If successful this study will support the concept of sit-stand desks as an effective long term school based intervention for benefits in health and learning in children across all demographics

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Any child with any disabilities that prevent them from standing up for short periods of time will be requested to continue with their usual practice of sitting at their school desk.
* Children with any disabilities or injuries/illnesses that prevent them from going about their usual routine will be excluded from the evaluation component of the intervention

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2015-08-20 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2016-07-15 (Actual)

PRIMARY OUTCOMES:
Sitting time (mins) | 7 days at baseline, 4 months, 8 months
  Change in time spent sitting using activPAL inclinometer device

SECONDARY OUTCOMES:
Standing time (mins) | 7 days at baseline, 4 months, 8 months
  Change in time spent standing using activPAL inclinometer device
Stepping time (mins) | 7 days at baseline, 4 months, 8 months
  Change in time spent stepping using activPAL inclinometer device
Steps | 7 days at baseline, 4 months, 8 months
  Change in Steps using activPAL inclinometer device
Sit to stand transitions | 7 days at baseline, 4 months, 8 months
  Change in Sit to stand transitions using activPAL inclinometer device
Total acceleration per minute | 7 days at baseline, 4 months, 8 months
  Change in Counts per minute using ActiGraph accelerometer device
Light physical activity (mins) | 7 days at baseline, 4 months, 8 months
  Change in Time spent in Light physical activity (mins) using ActiGraph accelerometer device
Moderate physical activity (mins) | 7 days at baseline, 4 months, 8 months
  Change in Time spent in Moderate physical activity using ActiGraph accelerometer device
Vigorous physical activity (mins) | 7 days at baseline, 4 months, 8 months
  Change in Time spent in vigorous physical activity using ActiGraph accelerometer device
Resting Systolic blood pressure (mmHg) | 7 days at baseline, 4 months, 8 months
  Change in Resting systolic blood pressure using automated Omron device
Resting diastolic blood pressure (mmHg) | 7 days at baseline, 4 months, 8 months
  Change in Resting diastolic blood pressure using automated Omron device
Height (m) | 7 days at baseline, 4 months, 8 months
  Change in height measured with portable Stadiometer
Weight (kg) | 7 days at baseline, 4 months, 8 months
  Change in weight measured with electronic weighing scales
Body Mass index (kg/m2) | 7 days at baseline, 4 months, 8 months
  Change in BMI calculated from height and weight measures
waist circumference (cm) | 7 days at baseline, 4 months, 8 months
  Change in waist circumference measured using anthropometry tape
Stroop test | 7 days at baseline, 4 months, 8 months
  Change in Computer based cognitive function test lasting 5 mins
Corsi block tapping test | 7 days at baseline, 4 months, 8 months
  Change in Computer based cognitive function test lasting 5 mins
Rapid visual information processing test | 7 days at baseline, 4 months, 8 months
  Change in Computer based cognitive function test lasting 5 mins
musculoskeletal discomfort | 7 days at baseline, 4 months, 8 months
  Change in discomfort using a self-report paper-based survey of 7 body parts. scale of 1-5, 1 is good, 5 is bad
Behaviour related mental health | 7 days at baseline, 4 months, 8 months
  Change in behaviour measured with a teacher completed 25 item Strengths and Difficulties questionnaire. each item is scored either "not true", "somewhat true" or "certainly true"

OTHER OUTCOMES:
Standing class fidelity | 30 minutes at 4 months
  sitting and standing behaviour recorded via direct observation by researcher
Experiences of using standing desks | 30 mins at 4 months
  focus groups with pupils exploring barriers and facilitators to sitting, standing and learning in the classroom
Experiences of teaching with standing desks | 60 mins at 4 months
  Interviews with teachers exploring barriers and facilitators to sitting, standing and teaching in the classroom

CONTACTS AND LOCATIONS:
Overall Officials: Stacy A Clemes, PhD, Principal Investigator — Loughborough University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sherry AP, Pearson N, Ridgers ND, Barber SE, Bingham DD, Nagy LC, Clemes SA. activPAL-measured sitting levels and patterns in 9-10 years old children from a UK city. J Public Health (Oxf). 2019 Dec 20;41(4):757-764. doi: 10.1093/pubmed/fdy181. PMID 30346570